CLINICAL TRIAL: NCT01160419
Title: Multicenter Study to Perioperative Chemotherapy for Resectable Adenocarcinoma in Gastric Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Prof. Dr. med. V. Heinemann, University of Munich - Klinikum Großhadern
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NEO-FLOT; EudraCT Nr.: 2008-007546-56
Record Dates: First submitted 2009-10-22; First posted 2010-07-12 (Estimated); Last update posted 2010-10-28 (Estimated); Status verified 2009-12

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — Docetaxel; Oxaliplatin; Leucovorin; Fluorouracil

ARMS (1):
- FLOT (Other): Docetaxel, Oxaliplatin, Folinic acid, 5-FU, q 2 weeks, application of 6 cycles
  Interventions: Drug: Docetaxel 50 mg/m2, 1-hour-Infusion, day 1; Drug: Oxaliplatin 85 mg/m², 2-hour-Infusion, day 1; Drug: Folinic acid 200 mg/m², 1-2-hour-Infusion, day 1; Drug: 5-FU 2600 mg/m², 24-hour-Infusion, day 1

INTERVENTIONS:
Drug: Docetaxel 50 mg/m2, 1-hour-Infusion, day 1 — 50 mg/m2, 1-hour-Infusion, day 1
Drug: Oxaliplatin 85 mg/m², 2-hour-Infusion, day 1 — 85 mg/m², 2-hour-Infusion, day 1
Drug: Folinic acid 200 mg/m², 1-2-hour-Infusion, day 1 — 200 mg/m², 1-2-hour-Infusion, day 1
Drug: 5-FU 2600 mg/m², 24-hour-Infusion, day 1 — 2600 mg/m², 24-hour-Infusion, day 1

SUMMARY:
The rationale of the NEO-FLOT-trial consists of an intensification of the neoadjuvant treatment.

This strategy is based upon the clear advantage of perioperative treatment and the fact, that in former trials adjuvant treatment could only be given in half of the patients (Cunningham 2006, Boige 2007).

In this study neoadjuvant chemotherapy is applied during a period of 12 weeks with an interim staging after 6 weeks.Due to the favourable efficacy and toxicity data the FLOT-regimen was chosen for the neoadjuvant treatment consisting of oxaliplatin, docetaxel, folinic acid and 5-Fluorouracil (Al-Batran 2008).

Postoperative treatment according to the results of the MAGIC trail is not part of the trail and is given at the responsibility of the participating centres.

ELIGIBILITY:
Inclusion Criteria:

* Histologically Confirmed Adenocarcinoma of the Gastroesophageal Junction (AEG I-III) or Gastric Adenocarcinoma (every T, N+ or T3/T4, Nx, M0)
* Written Informed Consent
* Age ≥ 18 Years
* Expected operability
* ECOG ≤ 2
* Exclusion of Peritoneal Metastasis
* Adequate Hematological, Renal, Cardiac and Hepatic Function
* Effective Contraception

Exclusion Criteria:

* Prior Chemotherapy or Radiotherapy of the Adenocarcinoma of the Gastroesophageal Junction (AEG I-III) or Gastric Adenocarcinoma
* Not Histologically Confirmed Primary Tumor
* Distant Metastasis, Local Relapse
* Known Hypersensitivity for 5-Fluorouracil, Leucovorin, Oxaliplatin or Docetaxel
* Known Dihydropyrimidin-Dehydrogenase (DPD) - Deficiency
* Peripheral Polyneuropathy ≥ Grade II (NCI-CTCAE, Version 3.0)
* Myocardial Infarction in the last 3 Months, Cardiac Insufficiency Grade II-IV (NYHA)
* Severe Comorbidity or Acute Infections
* Pregnancy or Breast Feeding
* Insufficient Contraception
* Participation in another Clinical Trial (Simultaneously or 30 Days Prior to Enrollment)
* Malignancy <5 years (except: Carcinoma In Situ of the Cervix Uteri or Adequately Treated Basalioma of the Skin)
* Lack of Legal Capacity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Estimated)
Dates: Start 2009-12; Primary Completion 2011-05 (Estimated); Study Completion 2014-05 (Estimated)

PRIMARY OUTCOMES:
Collection of the R0-Resection rate | 12 weeks
  after 6 cycles of biweekly FLOT chemotherapy and operation.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Munich, Klinikum Grosshadern, Munich, Germany